CLINICAL TRIAL: NCT02554110
Title: A Randomized Control Trial of the Oxistimulator as an Adjunct to Standard Practice to Decrease Extent and Duration of Oxygen Desaturation in Adult Patients Who Have Received Anesthetics or Are Receiving Sedating Medications
Brief Title: Peripheral Nerve Stimulation to Reduce Hypoxic Events
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Hugh M. Smith, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-003533
Record Dates: First submitted 2015-09-17; First posted 2015-09-18 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Apnea; Hypoventilation; Hypoxemia
MeSH Terms: conditions — Apnea; Hypoventilation; Hypoxia

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulator Active Device (Experimental): Intervention: This intervention arm will use a Stimulator Active Device peripheral nerve stimulation. Participants will receive a cutaneous stimuli in response to oxygen desaturations in postoperative surgical patients.
  Interventions: Device: Stimulator active device
- Stimulator Sham Device (Sham Comparator): No intervention: This arm will use a Stimulator Sham Device peripheral nerve stimulation.Participants will not receive a cutaneous stimuli in response to oxygen desaturations in postoperative surgical patients.
  Interventions: Device: Stimulator sham Device

INTERVENTIONS:
Device: Stimulator active device — This is a stimulator active device that delivers peripheral nerve stimulation in conjunction with pulse oximetry information.
  Arms: Stimulator Active Device
Device: Stimulator sham Device — This is an stimulator sham device that is not providing peripheral nerve stimulation.
  Arms: Stimulator Sham Device

SUMMARY:
This study is designed to determine if using peripheral nerve stimulation in conjunction with pulse oximetry as an adjunct to traditional monitoring in the PACU reduces the frequency and severity of sedation related apnea and hypoxic events.

DETAILED DESCRIPTION:
The primary effectiveness objective is to determine if transcutaneous stimulation will generate a respiratory response capable of reducing the extent and duration of oxygen desaturations in patients with presumed risk of obstructive sleep apnea (OSA) who have received some form of anesthesia or sedation. The primary safety objective is the demonstration that the peripheral nerve stimulation is safe for the use of preventing or reducing the sedation related hypoxemic events.

ELIGIBILITY:
Inclusion Criteria

* Males and females > 18 yrs old
* Flemon's Score > 15
* Able to provide written informed consent
* Having gynecological, colorectal, orthopedic surgery, and urologic surgeries
* Baseline oxygen saturation on room air > 96%

Exclusion Criteria:

* Peripheral neuropathy involving the upper extremities
* Procedures requiring direct admission to the ICU or any site other than the post-anesthesia care unit from the OR
* Diagnosed obstructive sleep apnea (OSA) and / or use of continuous positive airway pressure (CPAP) or biphasic positive airway pressure (BiPAP) in the PACU.
* Presence of any implantable electric devices, including internal defibrillators, pacemakers, or left ventricular assist device (LVAD)
* Post-procedure temperature < 35.5 Celsius or evidence of vasoconstriction
* Presence of metal hardware in either arm or in either shoulder
* Patients lacking access to the bare skin on an arm after surgery.
* History of atrial fibrillation
* History of bundle branch block
* Females from menarche to menopause that do not have a current negative pregnancy test or surgical history preventing pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-10-12 (Actual); Primary Completion 2017-01-19 (Actual); Study Completion 2017-01-19 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve for oxygen saturation (SpO2%) | One hour

SECONDARY OUTCOMES:
Frequency of desaturation episodes | One hour
Frequency of nursing interventions | One hour
Frequency of Adverse Events | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Smith, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith HM, Kilger J, Burkle CM, Schroeder DR, Gali B. Peripheral electrical stimulation reduces postoperative hypoxemia in patients at risk for obstructive sleep apnea: a randomized-controlled trial. Can J Anaesth. 2019 Nov;66(11):1296-1309. doi: 10.1007/s12630-019-01451-3. Epub 2019 Jul 23. PMID 31338807